CLINICAL TRIAL: NCT00651196
Title: Pilot Study - Type 1 Diabetes and Bone Health
Brief Title: Bone Health in Type 1 Diabetes
Acronym: DMB
Status: Completed | Type: Observational
Sponsor: Creighton University (Other)
Responsible Party: Principal Investigator, Laura Armas, Assistant Professor, Creighton University
Other Study IDs: Creighton5
Record Dates: First submitted 2008-03-30; First posted 2008-04-02 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-03

CONDITIONS: Type 1 Diabetes; Osteoporosis
Keywords: Type 1 diabetes; bone
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Osteoporosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Transilial bone specimens are retained for measurements
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Type 1 diabetics
- Healthy controls: Healthy age and sex matched controls

SUMMARY:
An increased skeletal fracture risk in diabetes has only recently been recognized. This human study is designed to elucidate the effect of Type 1 diabetes on bone remodeling and on structure.

DETAILED DESCRIPTION:
An increased skeletal fracture risk in diabetes has only recently been recognized. Human studies of patients with diabetes using bone mineral density and bone markers have noted low bone mass and mixed results on remodeling activity. Mouse models of diabetes have suggested that low bone turnover is the underlying problem. Low bone turnover could lead to an accumulation of microdamage that is not repaired causing compromised bone strength. Low bone turnover has not yet been confirmed in humans. This human study is designed to elucidate the effect of Type 1 diabetes on 1) bone remodeling, including histomorphometric and biochemical measures of bone formation and resorption, and 2) on structure, including micro architectural arrangement of trabeculae and bone mineral density.

ELIGIBILITY:
Inclusion Criteria:

* Age > 19 yrs or < 50 yrs.
* The diabetic subjects must have a diagnosis of Type 1 diabetes clinically defined as diabetes onset before age 50, acute presentation or diabetic ketoacidosis, with normal BMI. If history is equivocal, GAD antibodies > 1.45 U/mL will be used to define diagnosis.
* Diabetic subjects must be on insulin treatment.
* All subjects must have BMI between 18-30

Exclusion Criteria:

* On any medications that are known to interfere with bone metabolism including loop diuretics, steroids, anticonvulsants, bisphosphonates, metformin, glitazones
* Have normal or only mildly impaired kidney function defined as a calculated GFR greater than 60 mL/min/1.73m2
* History of cancer other than skin cancer
* Unstable angina, myocardial infarction, uncontrolled hypertension, malabsorption, active rheumatoid or collagen disease.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: males or females who are greater than 19 years of age and less than age 50 who have been diagnosed with type 1 diabetes for over 3 years.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
histomorphometry measurements | at 2nd visit

SECONDARY OUTCOMES:
peripheral QCT measurements | at 1st visit
micro CT measurements | at 2nd visit
nanoindentation measurements | at 2nd visit
Bone mineral density | at 1st visit

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Armas, MD, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States